CLINICAL TRIAL: NCT02787252
Title: Prospective, Clinical Pilot Study of High Frequency Wireless Spinal Cord Stimulation (SCS) in the Treatment of Chronic Pain With The Freedom Spinal Cord Stimulatory
Brief Title: Stimwave HF SCS Pilot Study
Acronym: HFSCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curonix LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30-00178
Record Dates: First submitted 2016-05-20; First posted 2016-06-01 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: FBSS
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HF DRG (Experimental): HF DRG Implants
  Interventions: Device: Implant procedure, Freedom Spinal Cord Stimulation System

INTERVENTIONS:
Device: Implant procedure, Freedom Spinal Cord Stimulation System — A needle is carefully inserted near the spinal cord. The stimulator is then slide through the needle to lay close to the spinal cord. The end of the stimulator is then sutured underneath the skin of the back.

SUMMARY:
The purpose of this study is to observe the efficacy of stimulation on over all pain relief as reported in an initial cohort of 6 patients treated with the Freedom High Frequency Spinal Cord Stimulator (SCS) System for low back and/or leg pain.

DETAILED DESCRIPTION:
This is a non-blinded, short-term study for a maximum duration of 12 weeks in which 6 patients will receive a Freedom SCS System. Subjects will have chronic, intractable pain of the trunk and/or lower limbs refractory to standard medical treatment; including unilateral or bilateral pain. Stimulators will be placed in the epidural space and over exiting nerve roots at vertebrae levels:

A. Bilateral T9-T10 epidural; B. Bilateral L1-L4 epidural. All Patients will be treated below perception threshold with High Frequency settings (10.000 Hz, 30 μs).

ELIGIBILITY:
1. Inclusion Criteria:

   A. Subject is ≥ 18 years of age at time of informed consent;

   B. Subjects have been diagnosed with chronic, intractable pain of the trunk and/or lower limbs with a VAS > 5cm (on a 10-cm scale);

   C. Subject diagnosis with chronic pain refractory to conventional medical management for at least 6 months prior to enrollment;

   D. Based on the medical opinion of the Principal Investigator, there is no evidence of anatomic abnormalities that could jeopardize the placement of the device or pose a hazard to the subject;

   E. Subject is willing to undergo surgical implant procedure, attend visits as scheduled, and comply with the study requirements;

   F. Based on the opinion of the Principal Investigator, subject is willing and able to operate the patient programmer, recharging equipment, diary and has the ability to undergo study assessments and provide accurate responses;

   G. Based on the opinion of the implanter, subject is a good surgical candidate for the implant procedure;

   H. Subject is male or non-pregnant female;

   I. Subject is deemed to be neuro-psycho-socially appropriate for implantation therapies based of the assessment of the investigator, using face-to-face encounters and the psychological testing described in the measures;

   J. Patient is capable of giving informed consent;

   K. Patient lives within reasonable distance from the study site (circumference of 75 km).
2. Exclusion Criteria:

A. Obvious mechanical instability related to pain (diagnosed by imaging taken within the past 6 months);

B. Malignancies;

C. Subject has post-herpetic neuralgia (shingles);

D. Subject has an active systemic infection or is immune-compromised.

E. Based on the medical opinion of the Principal Investigator the subject has other psychological conditions (e.g., psychosis, suicidal ideation, borderline personality disorder, somatization, narcissism), other health conditions (e.g., substance abuse, another chronic condition requiring the regular use of opioid medication), or other legal concerns that would preclude his/her enrollment in the study or potentially confound the results of the study;

F. Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study while participating in this study;

G. Insulin-dependent diabetic who is not controlled through diet and/or medication;

H. Bleeding complications or coagulopathy issues;

I. Pregnant/lactating or not using adequate birth control;

J. A life expectancy of less than one year;

K. Any active implanted device whether turned off or on;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Outcome (VAS) | 12 weeks post-implant
  The primary outcome is defined as the percentage of subjects who respond (50% average or more pain relief for back and leg pain) to SCS therapy at the end of 12 weeks post-implant of the system as compared to baseline with no increase in medication. The primary outcome will be measured with the VAS (100 mm line).
Primary Safety Outcome (Adverse Events) | 12 weeks post-implant
  Incidence and severity of device related adverse events during the study

SECONDARY OUTCOMES:
VAS | 12 weeks post-implant
  Percentage change from baseline in VAS for back and leg pain
ODI | 12 weeks post-implant
  Change from baseline in functionality using the ODI score

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Delta, Roeselare, West-Vlaanderen, Belgium